CLINICAL TRIAL: NCT05131737
Title: The Impact of Hypoxia on Patients With Precapillary Pulmonary Hypertension and Treatment of Adverse Effects
Brief Title: Exercise Endurance Time on the 2nd Day at 2500 m High Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: OVERALP II C
Record Dates: First submitted 2021-10-14; First posted 2021-11-23 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: High Altitude Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary edema of mountaineers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constant work-rate at altitude 2500 m above sea level (high altitude) (Experimental): Cycling at high altitude
  Interventions: Procedure: High altitude exposure; Procedure: Low altitude exposure
- Constant work-rate at altitude 470 m above sea level (low altitude) (Active Comparator): Cycling at low altitude
  Interventions: Procedure: High altitude exposure; Procedure: Low altitude exposure

INTERVENTIONS:
Procedure: High altitude exposure — Exposure to 2500m of altitude
Procedure: Low altitude exposure — Exposure to 490 m

SUMMARY:
The impact of a sojourn at 2500 m of high altitude for 26-30 h on constant work-rate exercise test time in patients with precapillary pulmonary hypertension

DETAILED DESCRIPTION:
Patients with pulmonary hypertension will perform a constant work-rate exercise test at low altitude (450m) and at high altitude 2500m in a randomized-cross-over sequence protocol. The constant work-rate exercise test time and other measures will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* PH class I (PAH) or IV (CTEPH) diagnosed according to guidelines: mean pulmonary artery pressure >20 mmHg, pulmonary vascular resistance ≥3 wood units, pulmonary arterial wedge pressure ≤15 mmHg during baseline measures at the diagnostic right-heart catheterization

Exclusion Criteria:

* resting partial pressure of oxygen <8 kilopascal at Zurich at 490 m low altitude
* exposure to an altitude >1000 m for ≥3 nights during the last 2 weeks before the study
* inability to follow the procedures of the study
* other clinically significant concomitant end-stage disease (e.g., renal failure, hepatic dysfunction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
cycle constant work-rate exercise test | 30 hours
  Difference in cycle constant work-rate exercise test (CWRET) time at 2500 vs. 490 m (Time Frame 24 to 30 hours)

SECONDARY OUTCOMES:
Heart rate | 30 hours
  Difference in cardiorespiratory measurements: Heart rate, during a cycle constant work-rate exercise test (CWRET) time at high altitude vs. low altitude
Ventilation in liters per minute | 30 hours
  Difference in cardiorespiratory measurements: Ventilation assessed in liters per minute, during a cycle constant work-rate exercise test (CWRET) time at high altitude vs. low altitude
Oxygen uptake | 30 hours
  Difference in cardiorespiratory measurements: oxygen uptake, during a cycle constant work-rate exercise test (CWRET) time at high altitude vs. low altitude
Oxygen saturation | 30 hours
  Difference in cardiorespiratory measurements: Oxygen saturation, during a cycle constant work-rate exercise test (CWRET) time at high altitude vs. low altitude
Partial pressure or oxygen | 30 hours
  Difference in partial pressure of oxygen at the beginning and end of a cycle constant work-rate exercise test (CWRET) time at high altitude vs. low altitude
Tricuspid pressure gradient | 30 hours
  Trans-tricuspid pressure gradient by echocardiography
Borg dyspnoea scale | 30 hours
  Difference in post-exercise Borg dyspnoea and leg fatigue scale during a cycle constant work-rate exercise test (CWRET) time at high altitude vs. low altitude
Visual analogue scale | 30 hours
  Difference in baseline in symptoms assessed by the Visual Analogue Scale at high altitude vs. low altitude
sit-to-stand test frequency | 30 hours
  Difference in baseline in sit-to-stand test frequency of standing up from a chair in a minute at high altitude vs. low altitude
6 minute walk test | 30 hours
  Difference in baseline in 6 minute walk test distance at high altitude vs. low altitude

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland